CLINICAL TRIAL: NCT04543435
Title: Investigation of Pain Coping Methods and Related Factors in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: European University of Lefke (Other)
Responsible Party: Sponsor
Other Study IDs: ÜEK/47/01/12/1920/05
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Pain
Keywords: postmenopausal; pain coping
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Musculoskeletal pain (MSP) reflects of musculoskeletal conditions related to tissues such as tendons, muscles, ligaments, nerves, and other joint structures. Coping strategies with pain are used to manage the pain and its impacts. The present study aimed to compare active and passive coping strategies used and pain severity in postmenopausal women according to their demographic characteristics. Also, the relationship between pain and coping strategies in postmenopausal women with cMSP will be examined.

DETAILED DESCRIPTION:
Musculoskeletal pain (MSP) reflects of musculoskeletal conditions related to tissues such as tendons, muscles, ligaments, nerves, and other joint structures. If MSP lasts for longer than three months, it becomes chronic. The prevalence of chronic MSP (cMSP) increases with aging and its ratio changes between 35,7% and 49,8%. The previous studies demonstrated the differences in the prevalence of cMSP between men and women. According to most of the studies, older women adults are more vulnerable to experience than men due to some differences in perception of pain such as biological characteristics, their roles in daily life, beliefs or coping strategies with pain.

Oestrogen has a prominent role in the physiology of muscles, tendons, ligaments, and bones. The decline of this sex hormone during menopause transition could lead to MSP, particularly in the postmenopausal period. Indeed, an increasing rate of cMSP in postmenopausal women has been reported.

Coping strategies with pain are used to manage the pain and its impacts. Coping with pain requires the self-regulation of individuals using cognitive and behavioral reactions. Dealing with cMSP is a process that can need the making of changes in daily life and activities This study aimed to compare active and passive coping strategies being used and pain severity in postmenopausal women according to their age, marital status, educational status, and exercise habits. Also, subdomains of strategies and subdomains of pain and the relationship between pain and coping strategies in postmenopausal women with cMSP will be examined.

ELIGIBILITY:
Inclusion Criteria:

* complaints of pain in anywhere of their body.
* presenting at least 1 year of amenorrhea
* being between the ages of 50-69 years.

Exclusion Criteria:

* have rheumatological, orthopedic and neurological diseases,
* have compression fractures, malignancies,
* have a chronic disease that will lead to secondary osteoporosis,
* have a drug use that will lead to secondary osteoporosis

Ages: 50 Years to 69 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women will be included.
Study Population: Patients presented to a rehabilitation clinic with complaints of pain in anywhere of their body and who are volunteer for the study will be included. Informed consent will be signed by the participants.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
McGill Pain Questionnaire | 15 minutes
  This tool is used for assesment of pain, namely; body part of pain, timeframe, characteristic and severity of pain. As score increases, pain condition worsens.
Pain Coping Inventory (PCI) | 10 minutes
  This tool is used for assessment of pain coping strategies. The higher score received means that coping strategy is used more.
Timed up and go test | 5 minutes
  This tool is used for assessment of functional mobility. The duration to complete the task (in seconds) is used as a score. As the score increase, the functional mobility decrease.

CONTACTS AND LOCATIONS:
Overall Officials: Beliz B Kaygısız, PT, PhD, Principal Investigator — European University of Lefke; Nuray Elibol, Study Director — Ege University; Sevim Acaröz Candan, Study Chair — Ordu University
Locations (1):
- European University of Lefke, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided